CLINICAL TRIAL: NCT04037306
Title: Measurements From Stool to Support Dietary Change
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Weight loss center programming suspended due to COVID-19 pandemic
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: Pro00094657
Record Dates: First submitted 2019-07-26; First posted 2019-07-30 (Actual); Last update posted 2020-09-02 (Actual); Status verified 2019-09

CONDITIONS: Diet Habit; Feeding Behavior; Behavior, Health
Keywords: Fiber
MeSH Terms: conditions — Feeding Behavior; Health Behavior

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rapid Feedback (Active Comparator): Participants received daily feedback on both fiber intake and stool butyrate measurements.
  Interventions: Behavioral: Butyrate Feedback; Behavioral: Fiber Feedback
- Delayed Feedback (Active Comparator): Participants received daily feedback on fiber intake and one-time feedback on stool butyrate measurements at the end of the study period.
  Interventions: Behavioral: Butyrate Feedback; Behavioral: Fiber Feedback

INTERVENTIONS:
Behavioral: Butyrate Feedback — Measure concentrations of stool butyrate by gas chromatography, returned to participants in summary report.
Behavioral: Fiber Feedback — Estimated fiber consumption from menu records of weight loss facility.

SUMMARY:
The purpose of the study is to evaluate if daily feedback on food-derived metabolites in stool enhances an individual's ability to make and/or sustain a dietary change.

DETAILED DESCRIPTION:
This is a research study to find out how people respond to information about food-derived compounds measured in their stool.

This study will take place over a three-week period. For these three weeks, participants in a medical weight loss program will be asked to collect samples of their stool daily from Monday to Friday, with optional sampling on weekends. We will measure the amount of butyrate, a breakdown product of fiber, in each sample provided and return this measurement by text message. Participants will be randomized into two groups: one group will have new measurements returned the day after providing each stool sample, and another will have their measurements returned all at once, at the end of the study. Both groups will also receive a daily text message report of their fiber intake, based on the foods they ordered at the weight loss facility cafeteria.

The greatest risks of the study include the possibility of infection while sampling stool, possible gastrointestinal discomfort from changes to the diet, and potential loss of confidentiality.

ELIGIBILITY:
Inclusion Criteria:

* between the ages of 18 and 80
* must be a client of the DFC (Duke Diet and Fitness Center) weight loss program for at least four continuous weeks.
* must have a smartphone

Exclusion Criteria:

* have diagnosis of Crohn's disease
* have known stricture (narrowing) of the intestine
* have any past history of intestinal obstruction

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2019-07-30 (Actual); Primary Completion 2020-03-10 (Actual); Study Completion 2020-03-10 (Actual)

PRIMARY OUTCOMES:
Change in nutrient intake, as estimated from menu selections | Baseline, Week 2, and Week 3
  Nutrient intake estimated in grams per day, summed over total menu selections.

SECONDARY OUTCOMES:
Change in butyrate concentration | Baseline, Week 2, and Week 3
  Butyrate measurements by gas chromatography, reported in mM (millimolar).

CONTACTS AND LOCATIONS:
Locations (1):
- Duke University Diet and Fitness Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No